CLINICAL TRIAL: NCT04998045
Title: Feasibility and Acceptability of a Peer-delivered Substance Use Screening and Brief Intervention for Youth Attending Rafiki Clinic in Eldoret, Kenya
Brief Title: Feasibility and Acceptability of a Substance Use Screening and Brief Intervention for Youth Living With HIV in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moi University (Other)
Collaborators: Indiana University (Other); Duke University (Other); Moi Teaching and Referral Hospital (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MoiU5; D43TW009345 (NIH)
Record Dates: First submitted 2021-06-26; First posted 2021-08-10 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Substance Use; Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Mass Screening; Crisis Intervention

STUDY DESIGN:
Intervention Model Description: All eligible youth will be screened for substance use and assigned to the intervention based on level of substance use risk. Immediately after the intervention they will rate the acceptability of the intervention. After enrollment is over, peers, clinic staff and youth will be asked to give feedback (qualitative and quantitative) on the feasibility and acceptability of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Youth aged 15-24 years Intervention: screening and brief intervention for substance use
  Interventions: Behavioral: Screening and brief intervention for substance use

INTERVENTIONS:
Behavioral: Screening and brief intervention for substance use — Screening will be done using the WHO Alcohol Smoking and Substance Involvement Screening Test (ASSIST). The brief intervention will be delivered based on ASSIST risk scores: low risk - verbal positive reinforcement and brief advice on harmful consequences of substance use (ii) moderate risk - brief motivational interviewing (BMI) (iii) high risk - BMI and referral to child psychiatry out-patient clinic. The BMI will be delivered in a single session (approximately 15 minutes) using Feedback Listen Options model (15): (i) providing feedback on screening results (ii) exploring pros and cons of substance use, enquiring about importance of change (iii) exploring options for change.

SUMMARY:
Youth living with HIV in Kenya frequently use substances and this negatively affects their mental health as well as viral suppression.

The goal of this study is to evaluate the feasibility and acceptability of a peer-delivered substance use screening and brief intervention for these youth.

DETAILED DESCRIPTION:
Globally, youth are disproportionately affected by substance use. In sub-Saharan Africa (SSA), an estimated 41% of youth have used at least one substance in their lifetime. Youth Living with HIV (YLH) have not been spared. In a study conducted in Kenya, 33% and 46% of youth attending a HIV clinic reported harmful patterns of alcohol and illicit substance use respectively. Substance use among YLH has been associated with negative outcomes including antiretroviral therapy (ART) non-adherence, neurocognitive deficits, poor virologic control and depression. Unfortunately, YLH in SSA lack access to substance use interventions. A study conducted by Parcesepe et al reported that only 37% of HIV adolescent sites in select LMICs offered any substance use screening and interventions.

The World Health Organization (WHO) recommends screening and brief intervention (SBI) in primary healthcare for identification and early intervention for substance use. Primary healthcare workers in LMICs are however often unable to implement SBI due to heavy workload. Peers represent a potential means through which SBI may be delivered in adolescent HIV settings and presents a number of advantages. First, peer support systems are well established in many adolescent HIV clinics in sub-Saharan Africa. Secondly, by drawing upon their shared experiences as youth living with HIV, the peers can provide empathic support to the adolescents.

Few studies have evaluated implementation of peer-delivered SBI for adolescents. Available studies have been conducted in high-income countries. To our knowledge, no study has evaluated implementation of peer-delivered SBI among YLH. Our project seeks to fill this gap by evaluating the feasibility and acceptability of a peer-delivered SBI for YLH in Kenya. This project is in line with: (i) Kenyan Ministry of Health guidelines for delivery of adolescent and youth friendly services which lists substance use counseling as an essential service, and (ii) United Nations Programme on HIV/AIDS (UNAIDS) Fast-track target 95-95-95, which requires that by 2030, 95% of people on ART be virally suppressed (12) as well as target 3.5 of the Sustainable Development Goals (SDGs) which requires that governments strengthen the treatment and prevention of substance abuse. Data from this study will set the stage for full-efficacy trials and ultimately to scale-up efforts to other LMICs.

ELIGIBILITY:
Inclusion criteria:

• Youth aged 15-24 years

Exclusion criteria

* those ill during the appointment
* those who decline to assent/consent
* youth unable to speak fluently in English.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Substance use assessed by the alcohol, smoking and substance involvement screening test (ASSIST) | baseline
  The ASSIST tool enquires about lifetime use of 9 substances (alcohol, tobacco, cannabis, cocaine, inhalants, amphetamines, opioids, hallucinogens and sedatives). Endorsement of lifetime use is followed by a series of questions enquiring about pattern of use in the past 3 months. Scoring for alcohol use is as follows: 0-10 Low; 11-26 Moderate; 27+ High. Scoring for all other substances is as follows: 0-3 Low; 4-26 Moderate; 27+ High

SECONDARY OUTCOMES:
level of depressive symptoms using the patient health questionnaire 9 | baseline
  It is a 9 item tool that examines for symptoms over the past two week period. Each of the 9 items is rated as follows: 0 - "not at all", 1 - "Several days", 2 - "More than half the days", 3 - "Nearly every day". Scoring: 0-4 minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-27 severe depression.
level of generalised anxiety using the 7 item generalised anxiety disorder scale | baseline
  It is a 7 item tool that examines for symptoms over the past two week period. Scoring: mild anxiety (5-9), moderate range (10-14), and severe range (15-21)
Fidelity to the intervention assessed using a researcher designed rating scale | during the intervention
  Fidelity checklists will be developed based on key elements of the intervention. Items will be rated by the SBI trainers on a 3-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: FLORENCE JAGUGA, MMED, Principal Investigator — MOI TEACHING & REFERRAL HOSPITAL
Locations (1):
- Florence Jaguga, Eldoret, RIFT Valley, Kenya

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the study after de-identification
Supporting Information: Study Protocol
Time Frame: immediately following publication no end date
Access Criteria: researchers whose proposed use of the data has been reviewed and approved by an IRB.

REFERENCES:
- [Background] Gamarel KE, Brown L, Kahler CW, Fernandez MI, Bruce D, Nichols S; Adolescent Medicine Trials Network for HIV/AIDS Intervention. Prevalence and correlates of substance use among youth living with HIV in clinical settings. Drug Alcohol Depend. 2016 Dec 1;169:11-18. doi: 10.1016/j.drugalcdep.2016.10.002. Epub 2016 Oct 11. PMID 27750182
- [Background] Gaitho D, Kumar M, Wamalwa D, Wambua GN, Nduati R. Understanding mental health difficulties and associated psychosocial outcomes in adolescents in the HIV clinic at Kenyatta National Hospital, Kenya. Ann Gen Psychiatry. 2018 Jul 10;17:29. doi: 10.1186/s12991-018-0200-8. eCollection 2018. PMID 30002721
- [Background] Parcesepe AM, Lancaster K, Edelman EJ, DeBoni R, Ross J, Atwoli L, Tlali M, Althoff K, Tine J, Duda SN, Wester CW, Nash D; IeDEA Consortium. Substance use service availability in HIV treatment programs: Data from the global IeDEA consortium, 2014-2015 and 2017. PLoS One. 2020 Aug 27;15(8):e0237772. doi: 10.1371/journal.pone.0237772. eCollection 2020. PMID 32853246
- [Background] Peltzer K, Matseke G, Azwihangwisi M. Evaluation of alcohol screening and brief intervention in routine practice of primary care nurses in Vhembe district, South Africa. Croat Med J. 2008 Jun;49(3):392-401. doi: 10.3325/cmj.2008.3.392. PMID 18581618
- [Background] Mark D, Hrapcak S, Ameyan W, Lovich R, Ronan A, Schmitz K, Hatane L. Peer Support for Adolescents and Young People Living with HIV in sub-Saharan Africa: Emerging Insights and a Methodological Agenda. Curr HIV/AIDS Rep. 2019 Dec;16(6):467-474. doi: 10.1007/s11904-019-00470-5. PMID 31776974
- [Background] Winn LAP, Paquette KL, Donegan LRW, Wilkey CM, Ferreira KN. Enhancing adolescent SBIRT with a peer-delivered intervention: An implementation study. J Subst Abuse Treat. 2019 Aug;103:14-22. doi: 10.1016/j.jsat.2019.05.009. Epub 2019 May 14. PMID 31229188
- [Background] Humeniuk R, Ali R, Babor TF, Farrell M, Formigoni ML, Jittiwutikarn J, de Lacerda RB, Ling W, Marsden J, Monteiro M, Nhiwatiwa S, Pal H, Poznyak V, Simon S. Validation of the Alcohol, Smoking And Substance Involvement Screening Test (ASSIST). Addiction. 2008 Jun;103(6):1039-47. doi: 10.1111/j.1360-0443.2007.02114.x. Epub 2008 Mar 28. PMID 18373724
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Musyoka CM, Mbwayo A, Donovan D, Mathai M. Alcohol and substance use among first-year students at the University of Nairobi, Kenya: Prevalence and patterns. PLoS One. 2020 Aug 28;15(8):e0238170. doi: 10.1371/journal.pone.0238170. eCollection 2020. PMID 32857791
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kohrt BA, Ramaiya MK, Rai S, Bhardwaj A, Jordans MJD. Development of a scoring system for non-specialist ratings of clinical competence in global mental health: a qualitative process evaluation of the Enhancing Assessment of Common Therapeutic Factors (ENACT) scale. Glob Ment Health (Camb). 2015;2:e23. doi: 10.1017/gmh.2015.21. Epub 2015 Dec 9. PMID 28593049
- [Derived] Jaguga F, Kwobah EK, Giusto A, Apondi E, Barasa J, Korir M, Rono W, Kosgei G, Puffer E, Ott M. Feasibility and acceptability of a peer provider delivered substance use screening and brief intervention program for youth in Kenya. BMC Public Health. 2023 Nov 16;23(1):2254. doi: 10.1186/s12889-023-17146-w. PMID 37974158